CLINICAL TRIAL: NCT02551913
Title: Effectiveness of Theory-based Sleep Hygiene Intervention in Improving Sleep Quality in Adolescents: a Cluster Randomized Controlled Trial
Brief Title: A Theory-based Sleep Intervention in Improving Sleep Quality in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Associate Professor and Director, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QUMS398
Record Dates: First submitted 2015-09-11; First posted 2015-09-16 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Sleep
Keywords: Psychological Theory; adolescents
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): The adolescents will not receive any specific information
  Interventions: Behavioral: Control
- Intervention (Experimental): The adolescents will receive relevant information on the importance of adequate sleep, the consequences of sleep deprivation, Provide information about others' approval,Provide normative information about others' behaviour,Goal setting ,action planning, coping planning, Set graded tasks,Prompt self-monitoring of sleep behaviour
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Control — the adolescents will not receive any specific intervention
  Arms: control
Behavioral: Intervention — A theory based sleep hygiene intervention based on the theory planned behavior will be conduced on the adolescent
  Arms: Intervention

SUMMARY:
Sleep education has been used as a method of primary and secondary prevention of sleep problems in all age groups. An especially vulnerable age group are adolescents who frequently have poor sleep habits and suffer from sleep deprivation. In adolescents, insufficient sleep, inadequate sleep quality, and irregular sleep patterns are associated with daytime sleepiness, negative moods, increased likelihood of stimulant use, higher levels of risk-taking behavior, poor school performance, and increased risk of unintentional injuries. As an US study has shown, sleepiness was the major causal factor in many traffic accidents and more than 50% of sleep-related crashes involved drivers aged 25 or younger. The study was aimed to evaluate the effectiveness of a theory-based sleep hygiene intervention in improving sleep quality in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* They are not involved in any sleep education program
* study at secondary schools in Qazvin city
* Ability to understand Persian language

Exclusion Criteria:

* Does not meet inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2841 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported Sleep hygiene behavior | changes from baseline , 1 month and 6 Months follow-up
  Sleep behavior will be assessed through self-report employing 24-h recall of the previous night's sleep
Changes in Sleep duration | changes from baseline , 1 month and 6 Months follow-up
  Sleep duration will be measured using the Pittsburgh Sleep Quality Index (PSIQ). The PSQI is a self-administered questionnaire to assess subjective sleep quality during the previous month (Buysse et al., 1989). The self-rated items of the PSQI generate seven component scores (range of subscale scores, 0-3): sleep quality; sleep latency; sleep duration; habitual sleep efficiency; sleep disturbance; use of sleeping medication; and daytime dysfunction.

SECONDARY OUTCOMES:
Changes in psychological predictors of sleep hygiene behavior (attitude, subjective norms intention, perceived behavioral control , Self-monitoring, action planning and coping planning) | changes from baseline , 1 month and 6 Months follow-up
  psychological predictors of sleep hygiene behavior were assessed using a using a self-reported measure. All items are rated on a Likert-type scale, ranging from 1 to 5.
Adolescent Sleep Hygiene Scale | changes from baseline , 1 month and 6 Months follow-up
General Health Questionnaire | changes from baseline , 1 month and 6 Months follow-up
  A self-administered questionnaire will be given to each participant, in which the PSQI-I, the Iranian version of the General Health Questionnaire 12 (GHQ12-I)
Pediatric Daytime Sleepiness Scale | changes from baseline , 1 month and 6 Months follow-up
Sleep Disturbances Scale for Children | changes from baseline , 1 month and 6 Months follow-up
Changes in health-related quality of life | changes from baseline , 1 month and 6 Months follow-up
  health-related quality of life will be measured using the Pediatric Quality of Life Inventory™ Short Form 15 Generic Core Scales.
Sleep knowledge questionnaire | changes from baseline , 1 month and 6 Months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- The Organization for Education, Qazvin, Iran

REFERENCES:
- [Derived] Lin CY, Strong C, Scott AJ, Brostrom A, Pakpour AH, Webb TL. A cluster randomized controlled trial of a theory-based sleep hygiene intervention for adolescents. Sleep. 2018 Nov 1;41(11). doi: 10.1093/sleep/zsy170. PMID 30423178